CLINICAL TRIAL: NCT00675519
Title: Effects of Brief Intervention for General Hospital Inpatients With Unhealthy Alcohol Use in Taiwan: A Randomized, Controlled Trial
Brief Title: An Evaluation of the Brief Interventional for Problem Drinkers Among Medical Inpatients
Acronym: BI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Shen-Ing,Liu, Senior Visiting Staff, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DOH93-TD-1050
Record Dates: First submitted 2008-04-28; First posted 2008-05-09 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Problem Drinking
Keywords: problem drinkers
MeSH Terms: conditions — Alcoholism | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BI (Experimental)
  Interventions: Behavioral: Motivational enhancement therapy

INTERVENTIONS:
Behavioral: Motivational enhancement therapy — Motivational enhancement therapy begins with the assumption that the responsibility and capacity for change lie within the client. The therapist begins by providing individualized feedback about the effects of the patient's drinking. Working closely together, therapist and patient explore the benefits of abstinence, review treatment options, and design a plan to implement treatment goals.

SUMMARY:
Compared with control participants at post-intervention follow-ups, unhealthy drinkers who receive the screening and brief intervention will (1) report reduced alcohol consumption among all patients, and (2) report reduced alcohol-related problems and health care utilization.

DETAILED DESCRIPTION:
Alcohol use is associated with a number of adverse health and economic effects. Problem drinking is associated with increased mortality rates and with premature mortality. As a result of these findings, the testing of the effectiveness of alcohol abuse prevention strategies has become an important national research priority. Secondary prevention of alcohol problems covers the methods used for early detection and treatment of people with excessive alcohol consumption. These preventive methods are referred to as brief interventions. Brief intervention is a short-term counseling strategy based on motivational enhancement therapy that concentrates on changing patient behavior and increasing patient compliance with therapy. It has been shown to be effective for helping socially stable problem drinkers to reduce or stop drinking, for motivating alcohol-dependent patients to enter long-term alcohol treatment, and for treating some alcohol-dependent patients for whom the goal is abstinence. The aims of this study are to examine the outcomes of a brief intervention to reduce alcohol consumption by problem drinkers among medical inpatients in general hospital setting. The study design is a randomized controlled clinical trial. Patients will be recruited from adult patients who are admitted to medical or surgical wards of a general hospital. All adult inpatients of a general hospital, aged 18 to 65 years, will be consecutively screened with the Alcohol Use Disorders Identification Test for identifying the problem drinkers. All patients who screen positive and who have signed a consent form will be contacted by a researcher and invited to participate in a face-to-face interview to determine their eligibility for the trial. The inclusion criteria are problems drinkers, defined as men who drank more than 21 units a week and women who drank more than 14 units a week. Patients will be excluded from participation in the study if they are younger than 18 years or older than 65 years, and have attended an alcohol treatment program in the last 3 months. Screened positives will then be interviewed using the instrument of SCAN to confirm the diagnosis of alcohol use disorders. The patients who fulfill the criteria will be randomized into one of the three following groups: (1) control group will be provided with routine inpatient usual care; (2) experimental group 1: physicians and nurses in charge will be informed of the results of alcohol consumption screening, in addition to providing routine inpatient usual care; (3) experimental group 2 will receive brief intervention, in addition to treatment protocols provided for experimental group 1. Brief intervention, offered twice by well-trained therapists, is 15-minute short-term individual consultation, giving alcohol health education, increasing their motivation to alcohol abstinence, teaching alcohol abstinence principle, and in order to ameliorate the over-drinking problems in these cases. The main outcome measures are alcohol use measures, which will be evaluated at 12-week after the study recruitment.

ELIGIBILITY:
Inclusion Criteria:

* men aged 18-65 admitted to medical or surgical wards in a medical center in Taipei;
* Unhealthy alcohol users defined as men who currently (past 3 months) drank risky amounts, > 168 g alcohol per week or usually drank more than 32 g/ occasion.
* Patients provide written informed consent

Exclusion Criteria:

* Psychotic disorders or symptoms, bipolar disorder, major suicide risk,
* serious medical illness, or currently being treated in psychiatric clinics/or alcohol treatment program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2004-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the number of drinks per week | 4-, 9- and 12-month

SECONDARY OUTCOMES:
included days abstinent, the number of heavy drinking episodes (> 5 drinks/ occasion); the proportions of patients with risky drinking (> 14 drinks per week) , heavier drinking (> 20 drinks per week), alcohol-related problems and health care utilization. | 4-, 9 and 12-month

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan